CLINICAL TRIAL: NCT03992196
Title: A Remote, Open-Label, Long-Term, Follow-up Study to Determine the Safety, Tolerability, and Efficacy of Rotigotine Transdermal System as Monotherapy in Adolescents With Restless Legs Syndrome
Brief Title: A Follow-up Study of Rotigotine Patch in Adolescent Subjects With Restless Legs Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision; Not a safety decision
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RL0007
Record Dates: First submitted 2019-06-17; First posted 2019-06-20 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-09

CONDITIONS: Restless Legs Syndrome
Keywords: RLS; Neupro; Rotigotine
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rotigotine (Experimental): Subjects will be initiated on 1 mg/24 h rotigotine and up-titrated to a maximum of 3 mg/24 h rotigotine, with the aim of achieving the individually optimized dosage. Dose adjustment of rotigotine is allowed at any time during the following Maintenance Period up to a maximum dose of 3 mg/24 h. At the end of the Maintenance Period, subjects will be down-titrated.
  Interventions: Drug: Rotigotine 1 mg/24 h; Drug: Rotigotine 2 mg/24 h; Drug: Rotigotine 3 mg/24 h

INTERVENTIONS:
Drug: Rotigotine 1 mg/24 h — Pharmaceutical Form: transdermal patch Route of administration: transdermal use Concentration: Application of rotigotine transdermal patch with 1 mg/24 h (5 cm^2 patch size).
  Other Names: Neupro
Drug: Rotigotine 2 mg/24 h — Pharmaceutical Form: transdermal patch Route of administration: transdermal use Concentration: Application of rotigotine transdermal patch with 2 mg/24 h (10 cm^2 patch size).
  Other Names: Neupro
Drug: Rotigotine 3 mg/24 h — Pharmaceutical Form: transdermal patch Route of administration: transdermal use Concentration: Application of rotigotine transdermal patch with 3 mg/24 h (15 cm^2 patch size).
  Other Names: Neupro

SUMMARY:
The purpose of this study is to assess the long-term safety, tolerability and the long-term efficacy of rotigotine treatment in adolescents with idiopathic Restless Legs Syndrome (RLS).

ELIGIBILITY:
Inclusion Criteria:

* Subject weighs >=40 kg
* Subject has completed at least one dose step in SP1006, a previous study of rotigotine in adolescents with Restless Legs Syndrome (RLS), without meeting withdrawal criteria
* Female subjects must be surgically incapable of childbearing, or effectively practicing an acceptable method of contraception (oral/parenteral/implantable hormonal contraceptives, intrauterine device, or barrier and spermicide). Abstinence is an acceptable method. Subjects must agree to use adequate contraception during the study and for 4 weeks after their final dose of study drug
* Subject is expected to benefit from participation, in the opinion of the investigator

Exclusion Criteria:

* Subject is experiencing an ongoing serious Adverse Event (SAE) that is assessed to be related to rotigotine by the investigator or Sponsor
* Subject has active suicidal ideation as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the "Since Last Visit" version of the electronic Columbia Suicide Severity Rating Scale (eC-SSRS) at the final evaluation visit of the previous rotigotine study (ie, Visit 10 of SP1006)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (1):
- Rl0007 101, Culver City, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.clinicalstudydatarequest.com and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if a determination is made that the data cannot be adequately anonymized.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.clinicalstudydatarequest.com and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in December 2019 and concluded prematurely in September 2022. Study participants entered this study from the parent rotigotine study in adolescents (SP1006) (NCT03728933).
Pre-assignment Details: 10 participants were screened and considered enrolled, but only 9 participants were treated. The 10th participant was lost to follow-up prior dosing and no Adverse events were reported for this participant. Participant Flow refers to the Enrolled Set.
Groups:
- No Treatment: Participant signed the informed consent form but never received any study medication during the study.
- Rotigotine Final Dose 2 mg/24 h: Participants in this arm were initiated on 1 milligram (mg)/24 hours (h) rotigotine and up-titrated to a maximum of 2 mg/24 h rotigotine and the same dose was continued throughout the 1 year Maintenance Period. Dose adjustment was allowed at any time during the Maintenance Period, based on the investigator's assessment. At the end of the Maintenance Period, participants were down-titrated.
- Rotigotine Final Dose 3 mg/24 h: Participants in this arm were initiated on 1 mg/24 h rotigotine and up-titrated to a maximum of 3 mg/24 h rotigotine and the same dose was continued throughout the 1 year Maintenance Period. Dose adjustment was allowed at any time during the Maintenance Period, based on the investigator's assessment. At the end of the Maintenance Period, participants were down-titrated.
Period: Enrollment
Arm/Group | No Treatment | Rotigotine Final Dose 2 mg/24 h | Rotigotine Final Dose 3 mg/24 h
Started | 1 | 2 | 7
Completed | 0 | 2 | 7
Not Completed | 1 | 0 | 0
Not completed — lost to follow-up prior dosing | 1 | 0 | 0
Period: Treatment
Arm/Group | No Treatment | Rotigotine Final Dose 2 mg/24 h | Rotigotine Final Dose 3 mg/24 h
Started | 0 | 2 | 7
Completed | 0 | 2 | 1
Not Completed | 0 | 0 | 6
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Poor drug compliance withdrawn by team and sponsor | 0 | 0 | 1
Not completed — Withdrawal due to non-compliance | 0 | 0 | 1
Not completed — PI's decision due to investigational medicinal product non-compliance | 0 | 0 | 1
Not completed — Withdrawal by parent/guardian | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Set consisted of all participants who had at least one patch (rotigotine) applied. Due to data protection/data privacy, data cannot be reported for a single participant.
Groups:
- Rotigotine Final Dose 2 mg/24 h: Participants in this arm were initiated on 1 mg/24 h rotigotine and up-titrated to a maximum of 2 mg/24 h rotigotine and the same dose was continued throughout the 1 year Maintenance Period. Dose adjustment was allowed at any time during the Maintenance Period, based on the investigator's assessment. At the end of the Maintenance Period, participants were down-titrated.
- Total: Total of all reporting groups
Arm/Group | Rotigotine Final Dose 2 mg/24 h | Rotigotine Final Dose 3 mg/24 h | Total
Number analyzed (Participants) | 2 | 7 | 9
Age, Customized [Count of Participants; unit: Participants]
  Adolescents (12-17 years) | 2 | 7 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 5 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 1
  White | 2 | 6 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. TEAEs were defined as events that started during the Treatment Period or within 30 days following the end of the Treatment Period (ie, on or after the date of first patch application and within 30 days following the date of last patch removal + 1 day), or those events where the intensity worsened within this time frame.
Time Frame: From Baseline until the Safety Follow-Up Visit (up to 14 Months)
Population: The Safety Set consisted of all participants who had at least one patch (rotigotine) applied.
Measure: Number; unit: percentage of participants
Arm/Group | Rotigotine Final Dose 2 mg/24 h | Rotigotine Final Dose 3 mg/24 h
Number analyzed (Participants) | 2 | 7
percentage of participants | 100 | 85.7

2. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Withdrawal of Study Medication
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. TEAEs were defined as events that started during the Treatment Period or within 30 days following the end of the Treatment Period (ie, on or after the date of first patch application and within 30 days following the date of last patch removal + 1 day), or those events where the intensity worsened within this time frame.
Time Frame: From Baseline until the Safety Follow-Up Visit (up to 14 Months)
Population: The Safety Set consisted of all participants who had at least one patch (rotigotine) applied.
Measure: Number; unit: percentage of participants
Arm/Group | Rotigotine Final Dose 2 mg/24 h | Rotigotine Final Dose 3 mg/24 h
Number analyzed (Participants) | 2 | 7
percentage of participants | 0 | 0

3. Secondary Outcome: Changes From Baseline in International Restless Legs Rating Scale (IRLS) Sum Score at Visit 9
Description: The IRLS consisted of 10 questions, each scored using a 5-point scale ranging from 0=not present to 4=very severe. The IRLS sum score was calculated by summing up the single scores of all applicable questions, i.e., the total sum score ranged from 0 (no RLS symptoms present) to 40 (maximum severity in all symptoms). A score between 31 and 40, indicates very severe RLS. A score between 21 and 30 indicates severe RLS. A score between 11 and 20 indicates moderate RLS. A score between 1 and 10 indicates mild RLS and a score of 0 means no RLS. A negative change from Baseline indicates improvement.
Time Frame: Visit 9 (Month 12), compared to Baseline (in SP1006)
Population: The Safety Set consisted of all participants who had at least one patch (rotigotine) applied. Here, Number of Participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rotigotine Final Dose 2 mg/24 h | Rotigotine Final Dose 3 mg/24 h
Number analyzed (Participants) | 2 | 2
score on a scale | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues. | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues.

4. Secondary Outcome: Changes From Baseline in Clinical Global Impressions (CGI) Item 1 at Visit 9
Description: The Clinical Global Impressions Item 1 (Severity of Illness) score ranges from 0 to 7 as follows: 0=not assessed, 1=normal, not ill at all, 2=borderline ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, 7=among the most extremely ill. The CGI Item 1 was completed during an interview between the participant and the investigator or designee. A negative change from Baseline indicates improvement.
Time Frame: Visit 9 (Month 12), compared to Baseline (in SP1006)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rotigotine Final Dose 2 mg/24 h | Rotigotine Final Dose 3 mg/24 h
Number analyzed (Participants) | 2 | 2
score on a scale | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues. | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues.

5. Secondary Outcome: Changes From Baseline in Restless Legs-6 Rating Scales (RLS-6) at Visit 9
Description: The RLS-6 Rating Scales was designed to assess the severity of RLS and consisted of 6 subscales. The subscales assessed severity of symptoms at the following times of the day/evening: falling asleep, during the night, during the day at rest, and during the day when engaged in daytime activities (not at rest). In addition, the subscales assessed satisfaction with sleep and severity of daytime tiredness/sleepiness. Scores for each of the 6 subscales ranged from 0 (completely satisfied) to 10 (completely dissatisfied). The change from baseline was derived for each of the subscales and reported in this outcome measure. A negative change from Baseline indicates improvement.
Time Frame: Visit 9 (Month 12), compared to Baseline (in SP1006)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rotigotine Final Dose 2 mg/24 h | Rotigotine Final Dose 3 mg/24 h
Number analyzed (Participants) | 2 | 2
score on a scale
  Satisfaction with sleep | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues. | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues.
  Severity: RLS symptoms at falling asleep | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues. | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues.
  Severity: RLS symptoms during the night | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues. | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues.
  Severity: RLS symptoms during the day - at rest | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues. | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues.
  Severity: RLS symptoms during the day-not at rest | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues. | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues.
  How tired or sleepy during the day | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues. | NA (NA) — Summary statistics are not reported for N<3 due to small sample size and participant identification issues.

ADVERSE EVENTS:
Time Frame: From Baseline until the Safety Follow-Up Visit (up to 14 Months)
Description: TEAEs were defined as events that started during the Treatment Period or within 30 days following the end of the Treatment Period (i.e., on or after the date of first patch application and within 30 days following the date of last patch removal + 1 day), or those events where the intensity worsened within this time frame. AEs are presented for 9 treated participants in the Safety Set. 1 participant was enrolled, but did not report any AEs and is therefore not included.
Arm/Group | Rotigotine Final Dose 2 mg/24 h | Rotigotine Final Dose 3 mg/24 h
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/7
Other Adverse Events (participants affected / at risk) | 2/2 | 6/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine Final Dose 2 mg/24 h (N=2) | Rotigotine Final Dose 3 mg/24 h (N=7)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (5)
Application site erythema (General disorders) | 2 (2) | 2 (2)
Application site rash (General disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT03992196/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT03992196/SAP_001.pdf